CLINICAL TRIAL: NCT03821441
Title: Trail To Evaluate the Immunity Duration of Different Sequential Immunization Schedules and Effectiveness for Bivalent Oral Poliomyelitis Vaccine Co-administered With IPV Booster Immunization for Poliovirus Vaccine
Brief Title: Trail To Evaluate the Immune Effects of Primary and Booster Immunizations With Poliovirus Vaccine
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Guangxi Center for Disease Control and Prevention (Other Government)
Responsible Party: Principal Investigator, Jingsi Yang, Director, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 201518502-C（bOPV-PRO-C）
Record Dates: First submitted 2019-01-03; First posted 2019-01-29 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2018-05

CONDITIONS: Poliomyelitis
Keywords: bOPV; IPV; Sequential immunization; Immunity Duration; Booster Immunization
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- bOPV(Candy) (Experimental): bOPV (Candy): bivalent oral attenuated live poliomyelitis vaccine against type 1 and type 3 in Dragee Candy (Human Diploid Cell) Produced by Institute of Medical Biology, Chinese Academy of Medical Sciences.
  1g/pill,10 pills/pach,one pill each time; each pill containing polio virus≥5.92 lgCCID50 including type1 polio virus≥5.8 lgCCID50，type 3 polio virus ≥5.3lgCCID50.
  Interventions: Biological: bOPV(Candy)
- bOPV(Liquid) (Experimental): bOPV (Liquid): bivalent oral attenuated live poliomyelitis vaccine against type 1 and type 3 (Human Diploid Cell) Produced by Institute of Medical Biology, Chinese Academy of Medical Sciences.
  0.5ml or 1.0ml each bottle;total content of polio virus≥7.12lgCCID50/ml，type1 polio virus≥7.0 lgCCID50/ml，type 3 polio virus ≥6.5lgCCID50/ml.(2 drops each person;be be equivalent to 0.1ml each person )
  Interventions: Biological: bOPV(Liquid)
- bOPV（liquid） (Experimental): bOPV(Liquid):Poliomyelitis (Live) Vaccine Type I Type III (Human Diploid Cell), Oral Produced by Beijing Tiantan Biological Products Co., Ltd. 1.0ml each bottle,2 drops each person(be be equivalent to 0.1ml each person).(total content of polio virus≥6.12lgCCID50，type1 polio virus≥6.0 lgCCID50，type 3 polio virus ≥5.5lgCCID50 in each 0.1 ml)
  Interventions: Biological: bOPV(Liquid)

INTERVENTIONS:
Biological: bOPV(Candy) — A single dose of 1 pill orally of bOPV to subjects aged 48 months who recieved bOPV (candy) produced by institute of Medical Biology, Chinese Academy of Medical Sciences in primary immunization.
  If bOPV(candy/liquid) is not available ,in order to protect the rights and interests of subjects ,the investigator can adjust other poliovirus vaccine such as IPV replace bOPV.
  Arms: bOPV(Candy)
Biological: bOPV(Liquid) — A single dose of 2 drops (0.1 ml) orally of bOPV to subjects aged 48 months who recieved bOPV (liquid) produced by institute of Medical Biology, Chinese Academy of Medical Sciences in primary immunization.
  If bOPV(candy/liquid) is not available,in order to protect the rights and interests of subjects ,the investigator can adjust other poliovirus vaccine such as IPV replace bOPV.
  Arms: bOPV(Liquid)
Biological: bOPV(Liquid) — A single dose of 2 drops (0.1 ml) orally of bOPV to subjects aged 48 months who received tOPV (liquid) produced by Beijing Tiantan Biological Products Co., Ltd. in primary immunization.
  If bOPV(candy/liquid) is not available,in order to protect the rights and interests of subjects ,the investigator can adjust other poliovirus vaccine such as IPV replace bOPV.
  Arms: bOPV（liquid）

SUMMARY:
Trail To Evaluate the Immunity Duration of healthy children who already took part in " The safety and immunogenicity by different sequential schedules of bOPV and bOPV in dragee candy with sIPV, a randomized, double blind, single center and parallel phase Ⅲ clinic trial was performed in Infants of two-month old in Guangxi Province, China" and continue to search for the effects of booster immunization.

DETAILED DESCRIPTION:
According to the requirement of the Strategy of Polio Eradication & Endgame Strategic Plan 2013-2018, bivalent oral attenuated live poliomyelitis vaccine against type 1 and 3 (bOPV) and inactivated poliomyelitis vaccine made by Sabin strain (sIPV) need to be used to eradiation both the wild poliovirus and vaccine-derived poliovirus. To evaluate the safety and immunogenicity by different sequential immunization schedules of bOPV and bOPV in dragee candy with sIPV,a randomized, double blind, single center and parallel phase Ⅲ clinic trial was performed in Guangxi Province in China. A total of 1200 infants at 2 months old were selected, and randomlydivided into 12 different groups (100 individuals were included in each group) administrated the vaccines at 0, 28, 56 days schedule.The detail of each group as following:1)1-dose cIPV + 2-dose bOPV (Candy); 2)1-dose sIPV + 2-dose bOPV (Candy); 3)2-dose cIPV + 1-dose bOPV (Candy); 4)2-dose sIPV + 1-dose bOPV (Candy); 5)2-dose cIPV + 1-dose tOPV (Candy); 6)2-dose sIPV + 1-dose tOPV (Candy); 7)1-dose cIPV + 2-dose bOPV (Liquid); 8)1-dose sIPV + 2-dose bOPV (Liquid); 9)2-dose cIPV + 1-dose bOPV (Liquid); 10)2-dose sIPV + 1-dose bOPV (Liquid); 11)2-dose cIPV + 1-dose tOPV (Liquid); 12)2-dose sIPV + 1-dose tOPV (Liquid).Blood Sample was collected before vaccination and one month after the third dose of vaccination. Neutralization antibody against type I, Type I and Type III poliomyelitis virus were detected to evaluate the seroprotection rates and antibody geometric mean concentrations. The fecal samples were collected to test viral shedding.The safety by different sequential schedule of the vaccines was also evaluated.This part of study have already been done in 2016.

To further evaluate the immunity duration of different sequential immunization schedules for bOPV and IPV ,more importantly,trying to research the effectiveness of bOPV booster immunization,the previous study will continue.

The detail of the research as following:

The subject, who have already receipted 3-dose polio vaccine for primary immunization in phase III clinical trail in Guangxi and with the result of the paired-serum, are recruited again.In order to research the immunity durability of primary immunizations of primary immunization(3 doses of immunization),blood samples are collected from the subject aged 24 months,36 months and 48 months separately.Neutralization antibody titers for against type I, Type I and Type III poliomyelitis virus are detected,moreover,the positive rate and antibody geometric mean titers are analyzed.

A single dose of bOPV（liquid/candy) will be given orally to subjects at the age of 48 months which can in support of the effectiveness research of booster immunization with bOPV. To protect the rights and interests of subjects,the investigator can use other poliovirus vaccine such as IPV instead when bOPV（liquid/candy）is not available.

The anticoagulant blood will be collected separatly at 48 months and the 28 days after booster immunization from subjects,which will be used to detect cellular immune response.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have already taken part in phase 3 clinical trail in Guangxi and were vaccinated 3-dose primary immunization with polio vaccines .Moreover，the results of the selected paired serum are required.
* 24 months old(calendar month).
* Guardians understand the contents and requirements of this trail , meanwhile, voluntarily joined this study with informed consents.
* Able to attend all scheduled visits and to comply with all trial procedures(including vaccinate and blood collection)

Exclusion Criteria:

* Any booster immunization with polio vaccine after finishing 3-dose primary immunizations research.
* Polio virus infection was demonstrated in laboratory experiment.
* Participation in another clinical trial at the same times.
* Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives or increase the risk of subjects,such as acute or chronic diseases 、some abnormal detected by lab,and so on.

Ages: 24 Months to 48 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1165 (Estimated)
Dates: Start 2018-01-04 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Positive rate of anti-poliovirus antibodies. | at aged 24 months
  To evaluate the effectiveness of bivalent oral attenuated live poliomyelitis vaccine against type 1 and type 3 (Human Diploid Cell) (candy/liquid) co-administered with co-administered IPV by neutralization assay. Defined ≥ 8 (1/dil) for anti-poliovirus as positive.These data is used to calculate positive rate of anti-poliovirus antibodies.When anti-poliovirus antibodies level ≥ 8 (1/dil),there is protective effect on subjects.
Positive rate of anti-poliovirus antibodies. | at aged 36 months
  To evaluate the effectiveness of bivalent oral attenuated live poliomyelitis vaccine against type 1 and type 3 (Human Diploid Cell) (candy/liquid) co-administered with co-administered IPV by neutralization assay. Defined ≥ 8 (1/dil) for anti-poliovirus as positive.These data is used to calculate positive rate of anti-poliovirus antibodies.When anti-poliovirus antibodies level ≥ 8 (1/dil),there is protective effect on subjects.
Positive rate of anti-poliovirus antibodies. | at aged 48 months
  To evaluate the effectiveness of bivalent oral attenuated live poliomyelitis vaccine against type 1 and type 3 (Human Diploid Cell) (candy/liquid) co-administered with co-administered IPV by neutralization assay. Defined ≥ 8 (1/dil) for anti-poliovirus as positive.These data is used to calculate positive rate of anti-poliovirus antibodies.When anti-poliovirus antibodies level ≥ 8 (1/dil),there is protective effect on subjects.

SECONDARY OUTCOMES:
The GMT and of positive rate anti-poliovirus antibodies in different age. | at aged 24、36、48 months
  In order to know the duration of anti-poliovirus antibodies level.We will use the neutralization assay to research the duration of anti-poliovirus antibodies types1, 2, and 3 induced by bivalent oral attenuated live poliomyelitis vaccine against type 1 and type 3 (Human Diploid Cell) (candy/liquid) co-administered with IPV.Using the method of neutralization assay. Defined ≥ 8 (1/dil) for anti-Poliovirus as positive.The data are used to analysis the GMT 、 positive rate of poliovirus antibodies.
The adverse reaction and event of polio vaccine occur in subjects | following 28 days after the boosting dose of bOPV
  Local and systemic adverse events were active collected in subjects after boosting dose of bOPV.
The GMT 、seroconversion rate of poliovirus antibodies after booster immunization. | at aged 48 months and 28 days after the boosting dose of bOPV
  In order to know the rationality of booster immunization and make sure dose the subject need a booster immunization and when is the best time.The investigator will give one dose boosting vaccine（bOPV）when the subject aged 48 months.The type of bOPV (liquid/candy) depends on what kind of vaccine the child had eaten in" Randomized, Double Blind, Single Center, Parallel Trial to Evaluate the Safety and Immunogenicity by Different Sequential Immunization Schedules of Bivalent Oral Poliomyelitis Vaccine Co-administered With IPV in Infants Aged 2 Months." Using the method of neutralization assay to detect the poliovirus antibodies，defined ≥ 8 (1/dil) for anti-Poliovirus as positive.The data are used to analysis the GMT 、seroconversion rate of poliovirus antibodies.
Cellular immunity situation in booster immunization | at aged 48 months and 28 days after the boosting dose of bOPV
  The anticoagulant blood will be collected separatly at 48 months and the 28 days after booster immunization from subjects,which will be used to detect cellular immune response. The blood were measured by flow cytometry,luminex or microarray,etc.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaojun Mo, Master, Principal Investigator — Guangxi Province Center for Diseases Control and Prevention
Locations (1):
- Guangxi Provincial Center for Diseases Control and Prevention, Nanning, Guangxi, China